CLINICAL TRIAL: NCT01028105
Title: Evaluation of the Prevalence of Methicillin Resistant Staphylococcus Aureus Colonization in Pre-Surgical Patients and Post-Operative Infection
Brief Title: Incidence and Relationship of Positive Preoperative Methicillin Resistant Staphylococcus Aureus (MRSA) Screens and Post-operative Infections
Acronym: MRSA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment did not reach power, therefore study was administratively closed in 2013
Sponsor: Inova Health Care Services (Other)
Collaborators: Cardinal Health (Industry)
Responsible Party: Principal Investigator, Cynthia Hack, Principal Investigator, Inova Health Care Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 08.003
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Methicillin-resistant Staphylococcus Aureus Infection
Keywords: Preoperative screening; MRSA; Incidence; Postoperative infection; Preoperative MRSA Screening Incidence; Postoperative MRSA Infection Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No MRSA screening, Group b (No Intervention): Standard of care
- MRSA screening, Group a (Other): MRSA preoperative screening
  Interventions: Other: Preoperative MRSA screening

INTERVENTIONS:
Other: Preoperative MRSA screening — MRSA preoperative screening and post operative infection rate, 30 days post operative
  Arms: MRSA screening, Group a

SUMMARY:
The purpose of this study is to evaluate the prevalence of pre-surgical patients who are MRSA carriers. From an evidence-based practice perspective, findings from this study can be considered in the evaluation of the hospital SOP mandating pre-surgical MRSA screening requirements for patients with scheduled surgeries.

The central hypothesis to be addressed in this study is whether the MRSA colonization and subsequent post-operative infection are the equivalent in these populations.

DETAILED DESCRIPTION:
Design and Methods: Subjects in this study of 975 pre-operative, scheduled surgical patients are in one of the three following groups:

* Group 1 (N=325): Allocation sample of surgical patients required to be MRSA screened per hospital SOP (including patients having a positive MRSA history, orthopedic surgery, undergoing dialysis, or transfer from another hospital, nursing home, skilled nursing facility, or jail).
* Group 2 (N=650): Randomized sample (1:1 ratio) of surgical patients not required to be MRSA screened per hospital SOP, to one of the following two groups:

  * 2a (N=325): MRSA screening; or
  * 2b (N=325): No MRSA screening. All subjects were followed for 30 days post-operatively to determine the incidence of post-operative infection. Treatment, diagnostic, and hospitalization data were collected for patients diagnosed with post-operative infection.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-surgical out patient at ILH
2. Surgical procedure scheduled at least 2 days before surgery
3. Surgery being done at ILH operating room
4. Provision of signed ICF

Exclusion Criteria:

1. Patient 18 years of age or older who is deemed by the hospital incapable of providing Informed Consent
2. Inability to communicate in the English language

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 975 (Actual)
Dates: Start 2008-02; Primary Completion 2011-01 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to compare the prevalence of MRSA colonization and its relationship to post-operative infection in patients who are currently pre-operatively MRSA screened per SOP to those who are not. | 30 days

SECONDARY OUTCOMES:
The secondary objective is to compare medical charges associated with diagnosis and treatment of post-operative infections for these groups using cost-effectiveness analysis. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Karen G Speroni, BSN, MHSA, PhD, Study Director — Inova Loudoun Hospital
Locations (2):
- United States (2):
  - Inova Health Care Services, Falls Church, Virginia
  - Inova Loudoun Hospital, Leesburg, Virginia